CLINICAL TRIAL: NCT00000498
Title: Control of Hypertension by Non-Pharmacologic Means
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 17; R01HL024999 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2000-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases | interventions — Diet, Sodium-Restricted; Diet, Reducing; Ethanol; Antihypertensive Agents

INTERVENTIONS:
Behavioral: diet, sodium-restricted
Behavioral: diet, reducing
Behavioral: alcohol restriction
Drug: antihypertensive agents

SUMMARY:
To determine whether blood pressure could be controlled by nutritional-hygienic, non-pharmacologic means in hypertensives treated with drugs in the Hypertension Detection and Follow-up Trial (HDFP).

DETAILED DESCRIPTION:
BACKGROUND:

In the 1970s, many studies had been conducted to control blood pressure in individuals maintained at normotensive levels by the use of weight control and sodium restriction without the concomitant use of anti-hypertensives. The associations between weight, sodium and blood pressure had been well established, but data on the relationship of intervention to blood pressure control had been less so.

DESIGN NARRATIVE:

Patients were randomly assigned to one of three groups. The 95 patients in Group I were advised to control weight, reduce sodium intake, modify dietary and alcohol intake and were removed from pharmacologic treatment. The 44 patients in Group II were removed from pharmacologic treatment, with no other intervention. The 48 patients in Group III were continued on pharmacologic treatment, with no other intervention. The primary endpoint was the proportion in Groups I and II with diastolic blood pressure less than or equal to 90 mm Hg in the absence of antihypertensive drugs. Secondary endpoints were average diastolic and systolic pressures.

The study completion date listed in this record was obtained from the CRISP legacy data.

ELIGIBILITY:
Men and women with controlled hypertension.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1980-04; Study Completion 1983-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Grimm — MOUNT SINAI HOSPITAL; Jeremiah Stamler — Northwestern University

REFERENCES:
- [Background] Stamler R, Stamler J, Grimm R, Dyer A, Gosch FC, Berman R, Elmer P, Fishman J, Van Heel N, Civinelli J, et al. Nonpharmacological control of hypertension. Prev Med. 1985 May;14(3):336-45. doi: 10.1016/0091-7435(85)90060-x. PMID 3903735
- [Background] Stamler R, Stamler J, Grimm R, Gosch FC, Elmer P, Dyer A, Berman R, Fishman J, Van Heel N, Civinelli J, et al. Nutritional therapy for high blood pressure. Final report of a four-year randomized controlled trial--the Hypertension Control Program. JAMA. 1987 Mar 20;257(11):1484-91. doi: 10.1001/jama.257.11.1484. PMID 3546747
- [Background] Dyer AR, Stamler R, Grimm R, Stamler J, Berman R, Gosch FC, Emidy LA, Elmer P, Fishman J, Van Heel N, et al. Do hypertensive patients have a different diurnal pattern of electrolyte excretion? Hypertension. 1987 Oct;10(4):417-24. doi: 10.1161/01.hyp.10.4.417. PMID 3653970
- [Background] Stamler R, Grimm RH Jr, Dyer AR, Talano JV, Prineas R, Crow R, Berman R, Gosch FC, Elmer P, Stamler J. Cardiac status after four years in a trial on nutritional therapy for high blood pressure. Arch Intern Med. 1989 Mar;149(3):661-5. PMID 2645845
- [Background] McDonald AM, Dyer AR, Liu K, Stamler R, Gosch FC, Grimm R, Berman R, Stamler J. Sodium, lithium-countertransport and blood pressure control by nutritional intervention in 'mild' hypertension. J Hypertens. 1988 Apr;6(4):283-91. PMID 2454254